CLINICAL TRIAL: NCT04831502
Title: A Phase 1, Open Label, Randomized, Single-Dose, Replicate Crossover Study to Determine the Bioavailability of the Tablet Formulation Relative to the Capsule Formulation of TAK-906 and the Effect of Food on the Pharmacokinetics of the Tablet Formulation in Healthy Subjects
Brief Title: Bioavailability and Food Effect Study of Two Formulations of TAK-906
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-906-1005
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — trazpiroben

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1: TAK 906 50 mg (Treatment A+Treatment B+Treatment A+Treatment B+Treatment C) (Experimental): Participants will receive TAK-906 50 milligram (mg) as Treatment A (TAK-906 capsule) and Treatment B (TAK-906 tablet) under fasted conditions and Treatment C (TAK-906 tablet) under fed conditions, orally, once on Day 1 of Periods 1 to 5. A washout interval of at least 3 days will be maintained between each Treatment Period.
  Interventions: Drug: TAK-906
- Sequence 2: TAK-906 50 mg (Treatment B+Treatment A+Treatment B+Treatment A+Treatment C) (Experimental): Participants will receive TAK-906 50 mg as Treatment B (TAK-906 tablet) and Treatment A (TAK-906 capsule) under fasted conditions and Treatment C (TAK-906 tablet) under fed conditions, orally, once on Day 1 of Periods 1 to 5. A washout interval of at least 3 days will be maintained between each Treatment Period.
  Interventions: Drug: TAK-906

INTERVENTIONS:
Drug: TAK-906 — TAK-906 Tablets.
Drug: TAK-906 — TAK-906 Capsules.

SUMMARY:
The aim of this study is to understand how TAK-906 tablets and capsules are processed by the body in healthy adults under fasting conditions and also how TAK-906 tablets are processed by the body when taken with a high fat high calorie breakfast compared to fasting.

This study will require participants to stay at the clinical research unit for about 3 weeks to be monitored after receiving TAK-906.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-906. This study will compare the pharmacokinetics (PK) of single oral dose of 50 mg tablet (test [Treatment B]) relative to single oral dose of 50 mg capsule (reference [Treatment A]) under fasted conditions. The study will also explore the effect of food on 50 mg tablet formulation (Treatment C: high-fat/high-calorie meal) on TAK-906 PK following tablet administration relative to the fasted state (Treatment B).

The study will enroll approximately 24 participants. Participants will be randomly assigned to 1 of the 2 treatment sequences.

This single-center trial will be conducted in the United States. The overall time to participate in this study is approximately 60 days. Participants will be followed up for up to 14 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Continuous nonsmoker who has not used nicotine-containing products for at least 3 months prior to the first dosing and throughout the study, based on participant self-reporting and urine cotinine test.
2. Body mass index (BMI) greater than or equal to (>=) 18.0 and less than (<) 30.0 kilogram per square meter (kg/m^2) at the screening.
3. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiograms (ECGs) performed at the screening visit and before administration of the initial dose of trial drug, as deemed by the investigator or designee.

Exclusion Criteria:

1. Presence of infectious diseases (example, Coronavirus disease-19 [COVID-19] and flu) at the time of screening or check-in.
2. Any history of major surgery that may affect absorption, metabolism or excretion of study drug (example, intestinal resections, hepatectomy, nephrectomy, cholecystectomy), and/or digestive organ resection (except appendectomy).
3. History of any illness that, in the opinion of the investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
5. Positive urine drug or alcohol results at screening or check-in.
6. Positive urine cotinine at screening.
7. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
8. QT interval corrected for heart rate using Frederica's equation (QTcF) is greater than (>) 450 milliseconds (msec) or ECG findings are deemed abnormal with clinical significance by the Investigator or designee at screening.
9. Estimated creatinine clearance <90 milliliter per minute (mL/min) at screening.
10. Unable to refrain from or anticipates the use of:

    o Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing and throughout the study. After first dosing, acetaminophen (up to 2 grams [g] per 24 hours) may be administered at the discretion of the investigator or designee; sponsor must be consulted prior to administering acetaminophen to a participants.
11. Has been on a diet incompatible with the on-study diet, in the opinion of the investigator or designee, within 30 days prior to the first dosing and throughout the study.
12. Is lactose intolerant or unable/unwilling to eat the high-fat, high-calorie breakfast.
13. Donation of blood or significant blood loss within 56 days prior to the first dosing.
14. Plasma donation within 7 days prior to the first dosing.
15. Participation in another clinical study within 30 days or 5 half-lives (whichever is longer) prior to the first dosing. The 30-day window or 5 half lives (whichever is longer) will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Ratio of AUClast: Area Under the Concentration-time Curve From Time 0 to the Last Quantifiable Concentration Following TAK-906 Tablet Relative to TAK-906 Capsule Administration Under Fasted State | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Geometric Mean Ratio of AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity Following TAK-906 Tablet Relative to TAK-906 Capsule Administration Under Fasted State | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Geometric Mean Ratio of Cmax: Maximum Observed Plasma Concentration Following TAK-906 Tablet Relative to TAK-906 Capsule Administration Under Fasted State | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose

SECONDARY OUTCOMES:
Number of Participants Reporting one or More Adverse Events (AEs) | Baseline up to 14 days after the last dose of study drug in Period 5 (Day 31)
Number of Participants Reporting one or More Serious Adverse Events (SAEs) | Baseline up to 14 days after the last dose of study drug in Period 5 (Day 31)
Geometric Mean Ratio of AUClast: Area Under the Concentration-time Curve From Time 0 to the Last Quantifiable Concentration Following TAK-906 Tablet in fed state Relative to TAK-906 Tablet in Fasted State | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Geometric Mean Ratio of AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity Following TAK-906 Tablet in fed state Relative to TAK-906 Tablet in Fasted State | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Geometric Mean Ratio of Cmax: Maximum Observed Plasma Concentration Following TAK-906 Tablet in fed state Relative to TAK-906 Tablet in Fasted State | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Cmax: Maximum Observed Plasma Concentration After Single Dose of TAK-906 | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Quantifiable After Single Dose of TAK-906 | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity After Single Dose of TAK-906 | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
AUC%extrap: Percent of AUCinf Extrapolated After Single Dose of TAK-906 | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Tmax: Time to Reach Maximum Plasma Concentration After Single Dose of TAK-906 | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Tlag: Lag Time to First Quantifiable Concentration After Single Dose of TAK-906 | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Kel: Apparent Terminal First Order Elimination Rate Constant After Single Dose of TAK-906 | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
CL/F: Apparent Plasma Clearance After Single Dose of TAK-906 | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Vz/F: Apparent Volume of Distribution During the Terminal Elimination Phase After Single Dose of TAK-906 | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
t½: Terminal Half-life After Single Dose of TAK-906 | Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/606d6617620b3b001e9dbb59